Athens, 1. 06. 2025

The effectiveness and efficacy of the combination of pharmacotherapy with the two new recovery-oriented programs, RECOVERTRSGR for patients with treatment- resistant schizophrenia and RECOVERYTRSBDGR for patients with

treatment- resistant bipolar disorder.

Dr. phil., Dipl.-Psych., Stavroula Rakitzi

Clinical psychologist and cognitive behavioral psychotherapist

Private practice

ILISION 34 15771 Athens Greece

2111180571

6989766935

Stavroula@Rakitzi.onmicrosoft.com

Description linkedin Stavroula Rakitzi

ORCID: http://0000-0002-5231-6619

Polyxeni Georgila, M. D. Psychiatrist and cognitive behavioral psychotherapist

Private practice

ILISION 34 15771 Athens Greece

6932905259

polyxenigeorgila@gmail.com

Description linkedin Polyxeni Georgila

ORCID: http://0000-0003-3137-506X

1

## Athens, 18/06/2025

## Informed consent to the research protocol

Dr. Stavroula Rakitzi, a clinical psychologist and cognitive behavioral psychotherapist, and Dr. Polyxeni Georgila, M.D., psychiatrist, will conduct research protocol regarding the effectiveness and efficacy of two newly developed programs, RECOVERYTRSGR for patients with treatment resistant schizophrenia and RECOVERYTRSBDGR for patients with treatment resistant bipolar disorder. RECOVERYTRSGR will be compared with treatment as usual (TAU) and RECOVERYTRSBDGR will be compared with treatment as usual (TAU). A randomization process after the baseline evaluation will be conducted in order to see which group you belong to.

These groups begin on 1.07. 2025 RECOVERYTRSGR has 190 sessions as well as the TAU group. RECOVERYTRSBDGR has 140 sessions as well as the TAU group. Both therapies aim to improve symptoms, cognitive functions, functional outcomes and recovery

The test results will be used for statistical analysis to research the effectiveness and efficacy of the treatments. Results will be anonymous, and no personal data will be displayed from any individual participating in the groups. I will let you know about the results. My participation in these groups is voluntary. I certify that I have been informed of the above and that I agree with them.

Athens, Name Signature